CLINICAL TRIAL: NCT03970746
Title: An Open-label, Dose-escalation, Phase I/II Study to Assess the Safety, the Tolerability, the Immunogenicity and the Preliminary Clinical Activity of the Therapeutic Cancer Vaccine, PDC*lung01, Associated or Not With Anti-PD-1 Treatment in Patients With Non-small-cell Lung Cancer (NSCLC)
Brief Title: Safety, Immunogenicity and Preliminary Clinical Activity Study of PDC*lung01 Cancer Vaccine in NSCLC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PDC*line Pharma SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PDC-LUNG-101; 2018-002382-19 (EudraCT Number)
Record Dates: First submitted 2019-05-17; First posted 2019-05-31 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Anti-PD-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A1 (Experimental): PDC*lung01 Low Dose
  Interventions: Biological: PDC*lung01; Drug: Alimta Injectable Product
- Cohort A2 (Experimental): PDC*lung01 High Dose
  Interventions: Biological: PDC*lung01; Drug: Alimta Injectable Product
- Cohort B1 (Experimental): PDC*lung01 Low Dose added to SoC, i.e., anti-PD-1 treatment
  Interventions: Biological: PDC*lung01; Drug: Keytruda Injectable Product
- Cohort B2 (Experimental): PDC*lung01 High Dose added to SoC, i.e., anti-PD-1 treatment
  Interventions: Biological: PDC*lung01; Drug: Keytruda Injectable Product

INTERVENTIONS:
Biological: PDC*lung01 — PDC*lung01 includes, in similar proportion, seven active agents, made of irradiated human plasmacytoid dendritic cells (PDC) loaded separately with a distinct synthetic peptide encoded by a lung tumor antigen, namely NY-ESO-1, MAGE-A3, MAGEA4, Multi-MAGE (an epitope common to several MAGE-A antigens), SURVIVN, MUC1 or a peptide derived from the Melan-A antigen.
Drug: Keytruda Injectable Product — The intention and decision to prescribe the anti-PD-1 monotherapy as SoC (TPS≥50%) must have been made by the investigator before and regardless of the patient's participation in the study.
  Other Names: Pembrolizumab
  Arms: Cohort B1; Cohort B2
Drug: Alimta Injectable Product — For patients with non-squamous NSCLC included in Cohorts A1 and A2, maintenance by pemetrexed (IV every 3 weeks) can be administered according to SoC.
  Other Names: Pemetrexed
  Arms: Cohort A1; Cohort A2

SUMMARY:
PDC-LUNG-101 trial is an open-label, dose-escalation, phase I/II study to assess the safety, the tolerability, the immunogenicity and the preliminary clinical activity of the therapeutic cancer vaccine, PDC*lung01, associated or not with anti-PD-1 treatment in patients with non-small-cell lung cancer.

DETAILED DESCRIPTION:
The therapeutic cancer vaccine, PDC*lung01 will be administered at two dose levels (low dose (LD) and high dose (HD)), as single agent or during maintenance treatment by pemetrexed (for adenocarcinomas in Cohorts A1 and A2) or added to the SoC (cohorts B1 and B2) i.e. anti-PD-1.

In cohorts A1 (low dose cohort) and A2 (high dose cohort), NSCLC patients will be treated at each of the six PDC*lung01 treatment visits with low dose/high dose administered successively by subcutaneous and then by intravenous route.

In cohort B1 and B2, the first PDC*lung01 injection will start within 48 hours after the first infusion of anti-PD-1. The fourth PDC*lung01 injection will occur within 48 hours after the infusion of the second cycle of anti-PD-1.

For each patient, the study will be divided into three consecutive parts:

* Pre-screening (for HLA-A*02:01 positivity), only patients with positive HLA-A*02:01 status will be proposed to be screened.
* Active period comprising a screening period, a treatment period (visits V1 to V6, during which the patient receives PDC*lung01 vaccine, at each visit), a V7 one week after the last injection and an end-of-treatment (EoT) visit (V8, 4 weeks after the last injection),
* Follow-up period which starts after the EoT visit and lasts up to two years after the first IMP administration.

ELIGIBILITY:
Inclusion criteria:

Pre-screening:

Documented HLA-A*02:01 positivity after the patient has provided written informed consent.

Only patients showing a documented positive result in pre-screening will be allowed to enter the screening period.

Screening:

1. Patients with histologically proven, or cytologically proven (allowed only for patients recruited in cohorts A1/A2), non-small-cell lung cancer (NSCLC). The stage of the disease is evaluated according to the classification of the American Joint Committee on Cancer, 8th edition (see Section 25.1)

   1. (i) Stage IIa/IIb/IIIa NSCLC following radical surgery (R0 resection) and, if applicable, following adjuvant platinum-based chemotherapy (Figure 2) -, or (ii) Stage IV histologically or cytologically confirmed case of epidermoid (squamous) lung cancer following 4 cycles of platinum-based therapy (Figure 3), if targeted treatment options were not indicated or (iii) Stage IV histologically or cytologically confirmed case of adenocarcinoma (non-squamous) lung cancer following 4 to 6 cycles of pemetrexed and platinum combination (Figure 3), if targeted treatment options were not indicated.

      (iv) Populations (ii) and (iii) who have stopped prematurely chemotherapy, after at least 2 cycles of platinum-based therapy, for any reason, AND do present with a documented stable disease or partial / complete response.
   2. For the anti-PD-1 immunotherapy (Cohorts B1 and B2):

      * The patient has first-line metastatic stage IV NSCLC measurable disease and is starting anti-PD-1. The intention and decision to prescribe the anti-PD-1 monotherapy as SoC (TPS≥50%), assuming no targeted mutation detected, following standard NGS testing, if applicable, and thus no targeted treatment option is indicated, must have been made by the investigator before and regardless of the patient's participation in the study. Radiotherapy/chemoradiotherapy for prior stage III NSCLC is allowed if the treatment-free interval is >1 year.
2. ECOG performance status 0 or 1.
3. Adequate renal and hepatic function as defined below:

   * Serum creatinine clearance > 50 mL/min (Cockcroft-Gault formula)
   * Bilirubin ≤ 1.5 times upper limit of normal (ULN)
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times ULN (up to 5 times ULN are allowed in case of presence of liver metastases).
4. Adequate haematological function as defined below:

   * Platelet count ≥ 70 x 10⁹/L;
   * White blood cell count ≥ 2.5 x 10⁹/L with
   * lymphocytes ≥ 1 x 10⁹/L, among which ≥ 10 % of CD8+ T cells at screening or at baseline and
   * absolute neutrophil count ≥ 1.5 x 10⁹/L;
   * Haemoglobin ≥ 90 g/L
5. Patient willing and able to provide a baseline blood sample for leucocyte enumeration, cellular allogeneic response and immune-monitoring of 100 ml in total (in one or two samplings).
6. For patients with brain metastases:

   * Central nervous system metastases are not symptomatic and have been treated,
   * In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤10mg daily prednisone (or equivalent) during at least 2 weeks before baseline.
7. For female patients without child-bearing potential: a documentation of tubal ligation or hysterectomy, ovariectomy or a post-menopausal status is available.

   For female patients of child-bearing potential: a negative serum pregnancy test at screening is required. The patient agrees to use a highly effective contraception method from signing informed consent form (screening), throughout the study treatment period with PDC*lung01 and for at least 28 days after the last administration of PDC*lung01.

   For female patients receiving Pemetrexed in cohorts A1/A2 concomitantly with PDC*lung01, according to corresponding SmPC, it is required to use effective contraception during treatment with pemetrexed.

   For female patients receiving Pembrolizumab in cohorts B1/B2 concomitantly with PDC*lung01, according to corresponding SmPC, it is required to use an effective method of contraception up to 4 months thereafter.

   A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

   A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

   "Highly effective" contraceptive measures acceptable for the whole duration of the study have been defined based on the CTFGs recommendations on contraception and are the following:
   1. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal),
   2. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable).
   3. Intrauterine device (IUD)
   4. Intrauterine hormone-releasing system (IUS)
   5. Monogamous relationship with a vasectomized partner. Partner must have been vasectomized for at least 6 months before the participant entered into the study
   6. Abstinence or absence of sexual relations with men.
8. Males with reproductive potential should use barrier method of contraception (condom) from signing informed consent form (screening) up to at least 28 days after the last dose of PDC*lung01.

   For male patients receiving Pemetrexed in cohorts A1/A2 concomitantly with PDC*lung01, according to corresponding SmPC, it is required to use barrier method of contraception up to 6 months thereafter.
9. In the Investigator's opinion, the patient is able and willing to comply with the requirements of the study.
10. Patient willing and able to sign the study informed consent form before any study-specific procedures are conducted.
11. Patient (male or female) is aged 18 years or above.
12. Specific for patients enrolled in France: Patient is affiliated to a health insurance system.

Exclusion criteria:

1. Mixed small-cell and non-small-cell histological features.
2. Patient has documented evidence of EGFR mutation, ALK fusion or ROS1 fusion (according to current ESMO clinical practice guidelines) or any mutation for which targeted treatment options would be indicated, as per SoC.
3. Patient has received immunotherapy or any investigational drugs within 4 weeks before the first PDC*lung01 dose. Chemoradiotherapy with consolidation durvalumab for prior stage III disease.
4. Patient with Stage IV disease that received prior radiotherapy (except palliative radiotherapy e.g. brain irradiation). Palliative radiotherapy for stage IV disease should be completed one week prior to baseline visit and for brain irradiation a 2-week window is required.
5. Patient without brain metastasis is receiving systemic corticosteroids at a dose level exceeding 10 mg/day (prednisone or equivalent) during the screening period (administration by nasal spray, topical solution or oral inhaler is non-systemic and is therefore allowed).
6. Patient has a medical history of cancer other than NSCLC, except the following: (i) non-melanoma skin cancer with complete resection, (ii) in situ carcinoma of the cervix, (iii) other cancer treated with no evidence of disease for at least five years.
7. Known hepatitis B and/or C infection (testing not required).
8. Known positive for human immunodeficiency virus (HIV; testing not required).
9. Uncontrolled congestive heart failure or hypertension, unstable heart disease (coronary artery disease with unstable angina or myocardial infarction within 6 months of baseline) or uncontrolled ventricular arrhythmias at the time of enrolment in the study (atrial fibrillation or flutter is acceptable).
10. Any history of splenectomy or splenic irradiation.
11. For female patients: pregnancy or lactation.
12. Any condition, including autoimmune or immunodeficiency active disease that, in the opinion of the Investigator, would jeopardise patient's safety, or might compromise the effect of the study drug or the assessment of the study result. Patients with vitiligo, diabetes Type I, psoriasis (not requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, or oral corticosteroids within the previous 12 months) or a history of autoimmune thyroiditis are not excluded.
13. Specific for patients enrolled in France: Patient is under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicities (DLT) related to the administration of PDC*lung01 | Up to one week after the last injection (Day 42)

SECONDARY OUTCOMES:
Occurrence of serious adverse events (SAEs) and adverse events (AEs), deemed as related to the association of PDC*lung01 and the anti-PD-1 therapy | Up to Day 63
Occurrence of serious adverse events (SAEs) and adverse events (AEs) | Up to Day 63
Detection of anti-HLA class I and II antibodies in the serum | Screening, Day 35 and Day 63
Ex vivo detection and characterization of CD8+ T cells against tumor antigens borne by PDC*lung01, using flow cytometry | Screening, Day 35 and Day 63
Objective Response Rate (according to RECIST version 1.1 for cohorts A1/A2 and iRECIST for cohorts B1/B2) | Day 63
Progression-Free Survival | 9 months from the first day of platinum-based or anti-PD-1 antibody administration

CONTACTS AND LOCATIONS:
Overall Officials: Johan Vansteenkiste, Prof, Principal Investigator — KU Leuven
Locations (16):
- Belgium (7):
  - Grand Hôpital de Charleroi, Charleroi
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - University Hospitals KU Leuven, Leuven
  - CHU Liège- Sart Tilman, Liège
  - AZ Delta vzw, Roeselare
  - AZ Sint-Nikolaas, Sint-Niklaas
- France (3):
  - CHU Grenoble, Grenoble
  - Centre Léon Bérard, Centre de lutte contre le cancer, Lyon
  - CHU Nantes, Nantes
- Germany (2):
  - Kliniken der Stadt Köln GmbH, Cologne
  - Universitätsklinikum Franlkfurt, Frankfurt am Main
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis - 's hertogenbosch, 's-Hertogenbosch
  - Antoni Van Leeuwenhoek (Nederlands Kanker Instituut), Amsterdam
  - Leiden University Medical Center (LUMC), Leiden
- University Clinical Centre, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PDC*line Pharma website — https://www.pdc-line-pharma.com/